CLINICAL TRIAL: NCT01637519
Title: Use of the PercSys MicroStent Device to Alleviate Ureteral Stone Symptoms and Hydronephrosis
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Percutaneous Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H11-00383
Record Dates: First submitted 2011-12-13; First posted 2012-07-11 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Kidney Stones
Keywords: kidney stones; ureteral stones; stent
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ureteral stone: Ten (10) patients with a unilateral, mid- or distal, ureteral (tube connecting kidney and bladder in the urinary system) stone will be enrolled and brought to completion in this study.

SUMMARY:
Kidney stones cause severe pain. Patients with a stone lodged in the ureter (the tube that drains the bladder), require urgent treatment with a stent to relieve the blockage. This tube, or ureteral stent, gives the patient relief until they can have their stone treated. This study is to evaluate a new type of ureteral stent to relieve pain from kidney stones. This stent is designed to drain the kidney and unlike other ureteral stents, is also designed to widen the ureter to help the stone pass on its own.

DETAILED DESCRIPTION:
This study is to evaluate a new type of ureteral stent to relieve kidney obstruction from a stone lodged in the ureter. This stent would be placed when a patient presents with pain in the Emergency Room or clinic in a patient that has no signs of infection. It is designed to continue drainage of the kidney and unlike other ureteral stents, is also designed to help dilate the ureter to facilitate spontaneous stone passage. This means the stent may also be therapeutic and the patient would be less likely to undergo another procedure to have the stone removed. Research performed at the Stone Centre at VGH shows that in ex vivo pig kidneys, this stent provides very good urinary drainage of the kidney. This has been published in a peer-reviewed journal (Lange D, Hoag NA, Poh BK, Chew BH. Drainage characteristics of the 3F MicroStent using a novel film occlusion anchoring mechanism. J Endourol. 2011 Jun;25(6):1051-6.).

ELIGIBILITY:
Inclusion Criteria:

1. Perforation of the urinary tract;
2. Acute hemorrhage;
3. Tissue trauma;
4. Edema;
5. Submucosal tunneling of guidewire or device during advancement; and
6. Protein encrustation of the device.

   Exclusion Criteria:
7. Infection;
8. Hemorrhage;
9. Complications associated with the use of anesthesia,
10. Perforation of the urethra or bladder,
11. Scarring or stricture of the urethra; and
12. Urinary retention due to urethral edema.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that present with a unilateral, mid- or distal, ureteral stone that require stent placement to relieve stone symptoms
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Relief of hydronephrosis (fluid in kidney causing kidney swelling) | 1-2 weeks following stent placement
  Patients will return for radiographic test(s) after the stent placement as determined by the physician which can include kidney-ureter-bladder (KUB) x-ray, renal and bladder ultrasound, or CT scan. This imaging helps determine 2 things: the degree of kidney swelling (hydronephrosis), stent migration and whether their stone is still present or not.

SECONDARY OUTCOMES:
Pain relief | 0, 1, 2, 3, 4, 5, 6, 7 post stent placement, and days 1 and 7 post stent removal
  Before stent placement the subject will complete Visual Analog Scale (VAS) questionnaire. After stent placement and discharge home study questionnaires will be completed each day at the end of the day, until stent removal which will be in approximately 7 days. Each VAS questionnaire takes approximately 10 minutes to complete. The subject will be instructed to bring these at their clinic visit for stent removal at Vancouver General Hospital. After the stent removal 2 more questionnaires are completed, at 1 day and at 7 days. These are sent back in a stamped return envelope.
Migration of stent | 1-2 weeks following stent placement
  Patients will return for radiographic test(s) after the stent placement as determined by the physician which can include kidney-ureter-bladder (KUB) x-ray, renal and bladder ultrasound, or CT scan. This imaging helps determine 2 things: the degree of kidney swelling (hydronephrosis), stent migration and whether their stone is still present or not.

CONTACTS AND LOCATIONS:
Overall Officials: Ben H Chew, MD, Principal Investigator — University of British Columbia, Vancouver General Hospital; Ryan F Paterson, MD, Study Director — University of British Columbia, Vancouver General Hospital
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Stone Centre, Vancouver General Hospital, Jim Pattison Pavilion, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No